CLINICAL TRIAL: NCT02349217
Title: Mindfulness Based Couples Therapy for Breast Cancer Survivors: A Pilot Study
Brief Title: Mindfulness Based Couples Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-0233; NCI-2015-00507 (Registry Identifier: NCI CTRP-Clinical Trials Reporting Registry)
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Breast cancer survivors; Breast cancer partners; Mindfulness-Based Relationship Enhancement; MBRE; Standard of care; Pain Assessment; Questionnaires; Surveys; Neurocognitive Tests; Cortisol Tests; Saliva tests; Interviews; Meditation; Yoga; Self-help materials
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires; Mental Status and Dementia Tests; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction Intervention (MBRE) (Experimental): Participant and partner take part in an 8-week Mindfulness-Based Relationship Enhancement (MBRE) intervention course. MBRE course consists of meditation and yoga techniques and handouts.
  Pain assessment administered at baseline and at follow up visit. Questionnaires completed at baseline and at follow up visit. Neurocognitive tests administered at baseline and at follow up visit. Cortisol testing performed after baseline visit and at follow up visit. Interviews conducted after follow up visit. These interviews are audio-taped and transcribed.
  Interventions: Behavioral: Mindfulness-Based Relationship Enhancement (MBRE); Behavioral: Pain Assessment; Behavioral: Questionnaires; Behavioral: Neurocognitive Tests; Procedure: Cortisol Tests; Behavioral: Interviews
- Standard of Care (Active Comparator): Participants receive self-help materials that have been previously developed by MD Anderson's Office of Public Education, the American Cancer Society, and the National Cancer Institute.
  Pain assessment administered at baseline and at follow up visit. Questionnaires completed at baseline and at follow up visit. Neurocognitive tests administered at baseline and at follow up visit. Cortisol testing performed after baseline visit and at follow up visit. Interviews conducted after follow up visit. These interviews are audio-taped and transcribed.
  Interventions: Behavioral: Self-Help Materials; Behavioral: Pain Assessment; Behavioral: Questionnaires; Behavioral: Neurocognitive Tests; Procedure: Cortisol Tests; Behavioral: Interviews

INTERVENTIONS:
Behavioral: Mindfulness-Based Relationship Enhancement (MBRE) — Participant and partner take part in an 8-week Mindfulness-Based Relationship Enhancement (MBRE) intervention course. MBRE course consists of meditation and yoga techniques and handouts.
  Arms: Mindfulness Based Stress Reduction Intervention (MBRE)
Behavioral: Self-Help Materials — Participants and partner receive self-help materials.
  Arms: Standard of Care
Behavioral: Pain Assessment — Pain assessment administered at baseline and at follow up visit. Pain assessment involves submerging hand in cold water.
Behavioral: Questionnaires — Questionnaires completed at baseline and at follow up visit. Questionnaires ask about fatigue, mood, stress, social support, marital satisfaction, depression, and general demographics (age, race and so on). It should take about 1½ hours total to complete the questionnaires.
  Other Names: Surveys
Behavioral: Neurocognitive Tests — Neurocognitive tests administered at baseline and at follow up visit. Tests to check memory and thinking abilities.
Procedure: Cortisol Tests — Cortisol testing performed after baseline visit and at follow up visit. Participants asked to collect saliva samples for cortisol assays immediately, 30, 45, and 60 minutes after awakening (representing the cortisol awakening response) and at noon, 4 P.M. and 8 P.M.
  Other Names: Saliva tests
Behavioral: Interviews — Interviews conducted after follow up visit. These interviews are audio-taped and transcribed.

SUMMARY:
The goal of this study is to explore the effects of a Mindfulness Based Couples Intervention on relationship satisfaction with quality of life and immune system function among breast cancer survivors and their partners.

DETAILED DESCRIPTION:
Baseline Visit:

If you are found to be eligible to take part in this research study, you will return to the clinic about a week later for the Baseline Visit. You will be instructed to fast (eat nothing and drink only water) for at least 8 hours before this visit.

* Blood (about 4-5 tablespoons) will be drawn for tests of your immune function, stress hormone levels, and blood sugar levels. After this blood test, you will be given breakfast.
* You will complete a pain assessment which involves you submerging your hand in cold water. Researchers will use your response to measure your pain tolerance.
* You will have electrocardiograms (EKGs) to check your heart function. The sensors will be attached at the beginning of the visit and then removed before you leave. You will be attached to the machine for several hours, but you will be able to be disconnected to take bathroom breaks, if needed.
* You will complete questionnaires about fatigue, mood, stress, social support, marital satisfaction, depression, and general demographics (age, race and so on). It should take about 1½ hours total to complete the questionnaires.
* You will complete a series of traditional neurocognitive tests (for example, tests to check your memory and thinking abilities). You will take these tests on the computer and with a pen and paper.
* Your blood pressure will be measured multiple times throughout the visit.

Study Groups and Interventions:

After the Baseline visit, you will be assigned to one of 2 groups. If you are in Group 1, you and your partner will take part in an 8-week Mindfulness-Based Relationship Enhancement (MBRE) intervention course designed to alleviate stress and other symptoms among couples. The MBRE course will consist of eight sessions taught by a professional Mindfulness instructor. The sessions will occur 1 time a week and last about 2½ hours each time. The MBRE course will consist of meditation and yoga techniques and handouts. The sessions will focus on teaching participants (all female breast cancer survivors and partners) the basics of Mindfulness Based Relationship Enhancement.

Attendance at these sessions and completion of daily homework assignments requiring up to 45 minutes per day are essential to the program.

If you are in Group 2, you will receive self-help materials that have been previously developed by MD Anderson's Office of Public Education, the American Cancer Society, and the National Cancer Institute.

Post-Intervention Follow-Up Visit:

If you are in Group 1, you will have a post-intervention follow-up visit about 12 weeks after your Baseline visit (4 weeks after you finish your 8-week intervention sessions). If you are in Group 2, you will have a post-intervention follow-up visit about 8 weeks after the Baseline Visit. You will fast for 8 hours before a post-intervention follow-up visit.

* Blood (about 4 to 5 tablespoons) will be drawn to check your immune function, stress hormone levels, and blood sugar. After the blood is drawn you will be given breakfast.
* You will complete the cold water pain tolerance test.
* You will have electrocardiograms (EKGs).
* You will complete questionnaires about fatigue, mood, stress, social support, marital satisfaction, depression, and general demographics (age, race and so on). It should take about 1½ hours total to complete the questionnaires.
* You will complete a series of traditional neurocognitive tests.
* Your blood pressure will be measured multiple times throughout the visit.

Cortisol Testing:

After the Baseline and Follow-up Visits, you will be asked to give samples to measure cortisol, a hormone related to stress. You will place a small cotton tube in your mouth for about 2 minutes, or until the swab is completely soaked with your saliva. After this, you will place the swab back in the tube, and freeze the sample. You will be given containers to hold the samples when you freeze them, as well as to mark which day and time each sample was collected. You will take these samples 7 times a day (right when you wake up; about 30, 45, and 60 minutes after waking; and then at noon, 4:00 p.m., and 8:00 p.m.). Researchers will use these samples to measure the changes in cortisol throughout the day. You will collect these samples for 2 days during the week, and 2 days on the weekend. After you complete 4 total days of collecting saliva samples after each visit, you will mail them back to MD Anderson in pre-paid envelopes.

Program Satisfaction Evaluations:

After the follow-up visits, the study staff will conduct individual interviews with a small group of participants. Interview questions will address participants' overall reactions to and satisfaction with the mind-body intervention, the impact they felt from social support, motivation, and their own ability for increasing physical activity and well-being. The study staff will also ask questions about both positive and negative effects of participating in the intervention. Interviews will be conducted by the PI or a trained research coordinator. All interviews will last no longer than 90 minutes and will be audio-taped using a digital recorder and transcribed. All audio files will be destroyed after they are transcribed.

This is an investigational study.

Up to 30 couples (60 participants) will take part in this research study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Stage 0-IIIA breast cancer survivors and their partner
2. All the female breast cancer survivors will be at least two months from receiving cancer treatment (surgery, adjuvant therapy or radiation) and within three years from completing cancer treatment, except for tamoxifen/aromatase inhibitors.
3. Are able to read and write in English
4. Are able to pass the Physical Activity Readiness Questionnaire or participant provides a letter from their physician or nurse practitioner clearing them for study participation
5. All couples co-habiting for at least 3 years with current partner who is willing to participate in study
6. Are 21 years of age or older

Exclusion Criteria:

1. Male breast cancer survivors;
2. Participants with a diagnosis of diabetes, unless they are able to provide a letter from a physician who will continue to monitor the participant during the research study
3. Anti-inflammatory medications (e.g. statins, cholesterol medication)
4. Consume excessive amounts of alcohol (>30 drinks/week)
5. Pregnant or thinking about becoming pregnant during the study period
6. Lactating women
7. Major medical conditions involving the immune system such as autoimmune and/or inflammatory diseases
8. Pressure readings >/=140/90 mm Hg, as defined by the 7th Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure, will be deemed ineligible to participate and excluded from the study. They will be referred to their family physician or community services. Those ineligible based on their initial blood pressure reading are allowed to participate if they provide a letter from a physician who will continue to monitor the participant during the research study.
9. A hemoglobin level < 10g/dl
10. Person less than 21 years of age

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01-23 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of Mindfulness Based Couples Therapy Intervention Among Breast Cancer Survivors and Their Partners (intervention adherence rate, defined as the proportion of sessions completed out of a total of 8 sessions) | 12 weeks
  Feasibility endpoint is intervention adherence rate, defined as the proportion of sessions completed out of a total of 8 sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dantzer, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org